CLINICAL TRIAL: NCT05147662
Title: A Phase 3, Single Group Treatment, Open-label, Study to Evaluate the Safety of BAY 94-9027 Infusions for Prophylaxis and Treatment of Bleeding in Previously Treated Children Aged 7 to <12 Years With Severe Hemophilia A
Brief Title: A Study to Learn How Safe the Study Treatment BAY94-9027 is and How it Affects the Body in Previously Treated Children Aged 7 to Less Than 12 Years With Severe Hemophilia A, a Genetic Bleeding Disorder That is Caused by the Lack of a Protein Called Clotting Factor 8 (FVIII) in the Blood
Acronym: Alfa-PROTECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21824; 2023-504388-18-00 (Registry Identifier: CTIS); 2021-004858-30 (EudraCT Number)
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Treatment of Bleeding; Prophylaxis of Bleeding; Hemophilia A; Children
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Main study (Part A) and the extension study (Part B) (Experimental): Part A will last for 6 months. After completing Part A participants will continue in the extension study for another 18 months.
  Interventions: Biological: Damoctocog alfa pegol (Jivi, BAY94-9027)

INTERVENTIONS:
Biological: Damoctocog alfa pegol (Jivi, BAY94-9027) — Part A: 40 IU/kg (up to 60 IU/kg at the investigator's discretion), two times per week (2x/week) with the first 4 infusions under medical supervision. Thereafter, participants will continue their treatment as home treatment. Dose may be increased up to 60 IU/kg if needed at any time during the study at the investigator's discretion.
  Part B: Each participant may continue on prophylaxis dose regimen as prescribed in part A (40 - 60 IU/kg, 2x per week) or adjustments to prophylaxis dose / dose frequency can be made at the investigator's discretion (based on the bleeding events and individual needs): Dose frequency may be decreased to every 5 days with a prophylaxis dose of 60 IU/kg.

SUMMARY:
Researchers are looking for a better way to treat hemophilia A. Hemophilia A is a genetic disorder where the body does not create enough of a protein called clotting factor 8 (FVIII) present in the blood. People with hemophilia A may bleed for a long time from minor wounds, have painful bleeding into joints, or have internal bleeding. In severe hemophilia A (clotting factor 8 levels less than 1%) bleedings are more likely to happen.

In this study researchers want to learn more about the treatment called BAY94-9027. BAY94-9027 is an injectable medicine used to replace missing clotting factor 8. In BAY94-9027 the clotting factor 8 has been pegylated (combined with a substance called polyethylene glycol (PEG)). This is to make the treatment last longer in the body so that less injections are required. BAY94-9027 is already available for the prevention and treatment of bleeding in adults and children who are 12 years and older. BAY 94-9027 is also called Jivi.

BAY94-9027 is not yet available for children aged 7 to less than 12 years. One potential specific risk of pegylated drugs is that proteins in the blood called antibodies are built. These may attach to the pegylation part of the drug and this in turn may lead to allergic reactions and the drug not working as well as it should during first 4 infusions. In studies that have been done so far, this has been seen in some children younger than six years, but not in 29 children aged 6 to less than 12 years treated with BAY94-9027. Further safety information related to how the body reacts to BAY94-9027 is however still needed for this age group.

The main purpose of this study is to learn how safe BAY94-9027 is (safety) and how it affects the body (tolerability) in previously treated children with severe hemophilia A who are between 7 to less than 12 years. To answer this question, the researchers will study information about two medical problems of special interest, if allergic reactions occur (also called hypersensitivity) and if the drug is not working as well as it should (also called loss of efficacy) during the first 4 infusions.

Allergic reactions may range from mild local reactions to widespread effects such as shortness of breath, skin rashes and low blood pressure. Only allergic reactions related to the study treatment will be considered.

The assessment if loss of efficacy occurred will be based on the occurrence of bleeding, the clotting factor 8 level in blood after injection called recovery, clotting factor 8 inhibitor tests and measurement of antibodies against the PEG.

The study has two parts, A and B. Part A takes 6 months and part B takes 18 months. In part A the participants will receive two injections of BAY94-9027 per week. In part B, the number of injections may be decreased, with up to five days between the injections. The participants in this study will visit the study site around 14 times and will have 15 phone visits. In part A, visit 1 is for screening. Visits 2 to 5 take place twice a week for two weeks. Visit 6 two weeks after visit 5, visits 7 to 10 take place monthly with visit 11 six weeks after visit 10. In part B, site visits will occur on month 9, 12, 18 and 24 and phone calls every month between the site visits. The participants' and their caregivers will record in an electronic patient diary information about when the study treatment was given and bleeding episodes that have happened.

During the study, the study doctors and their team will

* take blood samples,
* do physical examinations,
* review the participants' electronic diary
* ask questions about the participants' quality of life,
* ask the participants questions about how they are feeling and what adverse events they are having An adverse event is a medical problem that happens during the study. Doctors keep track of all adverse events that happen in study, even if they do not think the adverse events might be related to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participants with severe hemophilia A (participant's own FVIII activity [FVIII:C] <1%)
* Participants must be previously treated with FVIII concentrate(s) (plasma derived or recombinant) for a minimum of 50 exposure days (EDs) at the time of signing the informed consent
* Participant has understood the study if appropriate for his age, informed consent must be signed by the parent, the participant can only sign the assent
* Willingness and ability of participants and/or parents /caregivers to complete training in the use of the electronic patient diary (EPD) and to document infusions during the study

Exclusion Criteria:

* History of FVIII inhibitors
* Current evidence of inhibitor to FVIII measured using the Nijmegen-modified Bethesda assay (≥0.6 BU/mL) at the time of screening (central laboratory)
* Any other inherited or acquired bleeding disorder in addition to hemophilia A (e.g. von Willebrand disease, hemophilia B)
* Known hypersensitivity or allergic reaction to drug substance, excipients or mouse or hamster protein
* Any other significant medical condition that the investigator feels would be a risk to the patient or would impede the study
* Requires any pre-medication to tolerate FVIII treatment (e.g. antihistamines)
* Planned major surgery during the study
* Any individual who is receiving chemotherapy, immune modulatory drugs other than anti-retroviral chemotherapy, or chronic use of oral or intravenous (IV) corticosteroids (> 14 days) within the last 3 months
* Any individual who received commercially available subcutaneous factor substitution therapy (emicizumab) within the last 6 months
* The participant is currently participating in another investigational drug study or has participated in a clinical study involving an investigational drug within 30 days of study entry or previous participation in a clinical study with BAY94-9027

Ages: 7 Years to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2025-06-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- Arnold Palmer Hospital for Children, Orlando, Florida, United States
- Argentina (3):
  - Hospital de Niños Sor María Ludovica, La Plata, Buenos Aires
  - Instituo Hematología Arbesú, Godoy Cruz, Mendoza Province
  - Instituto de Hematología Dr. Rubén Dávoli, Rosario, Santa Fe Province
- Brazil (4):
  - HEMORIO, Rio de Janeiro, Rio de Janeiro
  - Hospital das Clínicas de Campinas - UNICAMP, Campinas, São Paulo
  - Hosp Clínicas Facult. Med. de Ribeirão Preto / USP, Ribeirão Preto, São Paulo
  - Irmandadade da Santa Casa de Misericordia de Sao Paulo (iSANTACASA), São Paulo, São Paulo
- McMaster Children's Hospital, Hamilton, Ontario, Canada
- Ospedale Pediatrico Bambino Gesù - Oncoematologia, Trapianto Emopoietico e Terapie Cellulari, Roma (RM), Lazio, Italy
- OUS Rikshospitalet Klinisk Forskningspost Barn, Oslo, Norway
- Turkey (Türkiye) (6):
  - Acibadem Adana Hastanesi, Çocuk Sagligi ve Hastaliklari, Çocuk Hematoloji-Onkoloji Bölümü, Adana
  - Hacettepe Üniversitesi Tip Fakültesi, Hacettepe Ihsan Dogramaci Çocuk Hastanesi,, Ankara
  - Akdeniz Üniversitesi Tip Fakültesi Çocuk Sagligi ve Hastaliklari Anabilim Dali Çocuk Hematoloji ve Onkoloji Bilim Dali, Antalya
  - Gaziantep Üniversitesi Tip Fakültesi, Sahinbey Arastirma Ve Uygulama Hastanesi, Çocuk Hematoloji ve Onkoloji Bilim Dali, Gaziantep
  - Ege Üniversitesi Tip Fakültesi, Çocuk Sagligi ve Hastaliklari Anabilim Dali, Çocuk Hematoloji Bilim Dali, Izmir
  - Ondokuz Mayis Üniversitesi Tip Fakültesi, Saglik Uygulama ve Arastirma Merkezi, Çocuk Sagligi ve Hastaliklari Anabilim Dali, Samsun

IPD SHARING:
Plan to Share IPD: No
There are no current plans to share data. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Ozelo MC, Luciani M, Glosli H, Kavakli K, Samji N, Makris GC, Tueckmantel C, Enriquez MM, Oliveira LC, Gupta S, Arbesu MG, Davoli M, Chan AKC, Mancuso ME. Plain Language Summary on Safety and Efficacy of Damoctocog Alfa Pegol in Previously Treated Children Aged 7 to < 12 Years With Severe Haemophilia A in the Phase 3, Open Label Alfa-PROTECT Main Study. Eur J Haematol. 2026 Jan 14. doi: 10.1111/ejh.70078. Online ahead of print. PMID 41531337
- [Derived] Ozelo MC, Luciani M, Glosli H, Kavakli K, Samji N, Makris GC, Tueckmantel C, Maas Enriquez M, Oliveira LC, Gupta S, Arbesu MG, Davoli M, Chan AKC, Mancuso ME. Safety and Efficacy of Damoctocog Alfa Pegol in Previously Treated Children Aged 7 to < 12 Years With Severe Haemophilia A in the Phase 3, Open Label Alfa-PROTECT Main Study. Eur J Haematol. 2026 Jan 4. doi: 10.1111/ejh.70059. Online ahead of print. PMID 41486550
- See also: Click here to find information on this study on Bayer's website. — https://clinicaltrials.bayer.com/study/21824
- Available data/document: CTIS Summary of Results: 2023-504388-18-00 — https://euclinicaltrials.eu/search-for-clinical-trials/?lang=en&EUCT=2023-504388-18-00
- Available data/document: Layperson Summary of Results: 2023-504388-18-00 — https://euclinicaltrials.eu/search-for-clinical-trials/?lang=en&EUCT=2023-504388-18-00

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 17 study centers in 7 countries between 23-Mar-2022 (first participant consent) and 04-Jan-2024 (last participant last visit in study part A).
Pre-assignment Details: Overall, 40 participants were screened. Of the 40 screened participants, 3 (7.5%) failed screening and 1 (2.5%) was not enrolled for other reasons. 36 (90%) participants were assigned to treatment and 35 (88%) participants received study treatment.
  These initial results comprise a 6-month treatment phase (Part A) with a minimum of 50 exposure days. Results for the subsequent 18-month extension (Part B) will be reported as part of the final results.
Groups:
- All Participants: All participants
Period: Overall Study
Arm/Group | All Participants
Started (Assigned to treatment) | 36
Treated (Received at least 1 dose of study treatment) | 35
Completed (Completed study part A) | 32
Not Completed | 4
Not completed — Withdrawal by parent/guardian | 3
Not completed — Assigned to treatment but never treated | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set A: participants enrolled into the part A of the study who had taken at least 1 dose of the study intervention.
Arm/Group | All Participants
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.63 (1.37)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 33
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events of Special Interest (AESI) Hypersensitivity and Loss of Efficacy Associated With the First 4 Exposure Days (EDs) Leading to Discontinuation
Description: The occurrence of the defined adverse events of special interest was documented during the first 4 days that a participant was exposed to the study intervention.
Time Frame: Individual first 4 exposure days
Population: The primary endpoint analysis was performed on the modified safety analysis set (n=34). One participant in the safety analysis set (which consisted of all participants enrolled into part A of the study who had taken at least 1 dose of the study intervention; n=35) was excluded from the primary endpoint assessment due to treatment discontinuation for any reason other than AESI before the 4th ED.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 34
Participants | 1

2. Secondary Outcome: Adverse Drug Reactions (ADRs)
Description: Adverse drug reactions were defined as any adverse events where a causal relationship of at least possibly related with the use of BAY 94-9027 had been ascribed by the investigator. In this study, treatment emergent study drug-related adverse events were used in defining ADRs.
Time Frame: Up to 24 months
Reporting Status: Not Posted, anticipated posting 2026-05

3. Secondary Outcome: Anti-drug Antibody (ADA) Development
Description: All participants were tested for the development of anti-drug antibodies (ADAs) (anti-polyethylene glycol [PEG] and anti-PEG immunoglobulin M [IgM]).
Time Frame: Up to 24 months
Reporting Status: Not Posted, anticipated posting 2026-05

4. Secondary Outcome: The Number of Participants With Confirmed Factor VIII Inhibitors
Description: A positive FVIII inhibitor test was defined with a threshold of ≥ 0.6 BU/mL at the central laboratory. The first positive measurement was confirmed by a second, different sample.
Time Frame: Up to 24 months
Reporting Status: Not Posted, anticipated posting 2026-05

5. Secondary Outcome: Annualized Bleeding Rate (ABR)
Description: For each participant, the number of bleeds was related to the individual observation period to assess bleeding rates. For descriptive analyses, bleeding rates were annualized at the individual participant level using the formula: ABR = (number of bleeds × 365.25 × 24 × 60)/(Period). Period was defined as the number of minutes calculated from the date and time of the beginning of the treatment period and the date and time of the end of the treatment period of interest.
Time Frame: Up to 24 months
Reporting Status: Not Posted, anticipated posting 2026-05

6. Secondary Outcome: BAY94-9027 Consumption
Description: Summary statistics for BAY 94-9027 consumption are provided for prophylaxis treatment, for treatment of bleeds, and overall. Consumption per year and per infusion is presented based on total dose (IU) and dose per body weight (IU/kg).
Time Frame: Up to 24 months
Reporting Status: Not Posted, anticipated posting 2026-05

7. Secondary Outcome: Number of Infusions/Month and Year (Annualized Infusion Rate)
Description: Number of infusions per month and year
Time Frame: Up to 24 months
Reporting Status: Not Posted, anticipated posting 2026-05

ADVERSE EVENTS:
Time Frame: From start of study intervention up to 26 weeks, with a mean and median duration of study intervention of 182 days at the time of interim analysis.
Description: Adverse event reporting for all-cause mortality considers all deaths that occurred at any time during the study before the last contact for interim analysis, from up to 30 days before start of study intervention until a mean and median duration on study intervention of 182 days at the time of these interim results, for a mean total of 182-212 days.
Groups:
- Prophylaxis: Prophylaxis
Arm/Group | Prophylaxis
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 1/35
Other Adverse Events (participants affected / at risk) | 20/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylaxis (N=35)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylaxis (N=35)
Vomiting (Gastrointestinal disorders) | 1 (1)
Injection site pruritus (General disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1)
Eye irritation (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Drug ineffective (General disorders) | 1 (1)
Injection site rash (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Infusion site pain (General disorders) | 1 (3)
Hypersensitivity (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 2 (2)
Otitis externa (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Viral pharyngitis (Infections and infestations) | 2 (2)
Periorbital cellulitis (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Respiratory sinus arrhythmia magnitude (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (5)
Seizure (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size is a limitation in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications before submission for publication and embargo such communications for 45 days. If confidential information is present, the sponsor can embargo proposed publications for an additional 75 days to seek protection of intellectual property. For multi-center studies, publication of results specific to the PI's institution can be embargoed for as long as a multi-center publication is not published, up to a maximum of 18 months.

DOCUMENTS (2):
  • Study Protocol (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT05147662/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT05147662/SAP_001.pdf